CLINICAL TRIAL: NCT03328611
Title: MCJR Joint Replacement Clinical Outcomes Database
Status: Recruiting | Type: Observational
Sponsor: Midwest Center for Joint Replacement (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: OMB No. 0990-0279
Record Dates: First submitted 2017-10-24; First posted 2017-11-01 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Joint Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Hip and Knee Joint Replacement — Hip and Knee Joint Replacement

SUMMARY:
The purpose of this research study is to develop a database of information regarding the diagnosis, treatment, and outcome of participants who have had a joint replacement. The more information gathered, the better the investigators will be able to treat future patients who need a joint replacement. For example the investigators learn what works well to help design implants and treatment protocols for the future. The investigators publish manuscripts and present research findings around the world to help other investigators and clinicians learn what is discovered. Furthermore, implant manufacturers may be able to use this information in the database to evaluate the success rates of specific joint replacement products.

DETAILED DESCRIPTION:
As part of our growing clinical tracking EMR system the investigators plan to collect preoperative and postoperative Patient Reported Outcome Measures (PROMS) on all patients with degenerative hip and knee disease. The investigators will collect PROMS along with implant device specific revision rates. This will be used for implant surveillance, clinical outcome tracking, return to work outcome metrics and failure modes and rates of various hip and knee implants. Information generated during regular hospital and clinic visits will be entered into the database. For example, x-ray findings done before surgery will be entered into the database. Surgery information will be entered into the database. The investigators will also enter demographic information into the database such as name, email, birthdate, gender, height, and weight. Medical co-morbidities such as diabetes, high blood pressure, and prior surgeries will also be entered.

The investigators will collect this information before surgery, during the operation, and at annual follow-up visits. The investigators will also contact patients via email with short outcome score surveys (known as Patient Reported Outcome Measures or PROM's). This will save many hours of return visits if scores indicate the joint replacements are doing well. Also this will trigger additional follow-up measures if PROMS scores drop off.

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of degenerative joint disease requiring treatment with a joint replacement

Exclusion Criteria: Clinical diagnosis of degenerative joint disease not requiring treatment with a joint replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Joint Replacement Patients: Clinical diagnosis of degenerative joint disease requiring treatment with a joint replacement of the hip and knee
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score | Change in OKS from Baseline at 1 year, assessed up to 30 years
  OKS - PROM
HOOS | Change in HOOS from Baseline at 1 year, assessed up to 30 years
  Hip Outcome scores
KOOS | Change in HOOS from Baseline at 1 year, assessed up to 30 years
  Knee Outcome scores

SECONDARY OUTCOMES:
radiographic findings | Change in radiographic findings from Baseline at 1 year, assessed up to 30 years
  x-ray reports of joint replacements

CONTACTS AND LOCATIONS:
Locations (1):
- Midwest Center for Joint Replacement, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Only de-indentified or anonymous data will be shared with other researchers through HIPPA compliant server.